CLINICAL TRIAL: NCT03652389
Title: i-Matter: Investigating an mHealth Texting Tool for Embedding Patient-reported Data Into Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-01044
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MJS DIABETES (Experimental): will receive and respond to daily PROs via ttext messages and report SMBG (if insulin-dependent) over the course of the 12-month study.
  Interventions: Behavioral: MJS Diabetes
- Usual Care (No Intervention): Standard Diabetes Treatment

INTERVENTIONS:
Behavioral: MJS Diabetes — patients will receive and respond to daily PRO (patient recorded outcomes) via text messages and report SMBG (self monitoring blood glucose), if insulin dependent, over the course of a 12 month period. They will also receive feedback and motivational messages based on patterns of their PROs
  Arms: MJS DIABETES

SUMMARY:
This study will integrate a technology-based patient-reported outcome (PRO) system [herein MJS DIABETES] that incorporates patients' perspective of their disease and functional status into the management of type 2 diabetes (T2D) in primary care practices. MJS DIABETES is an innovative mobile platform that utilizes text-messaging to capture patients' self-reported PROs in real-time; enhance patient engagement through data-driven feedback and motivational messages; and create dynamic visualizations of the PROs that can be shared in printed reports, and integrated into the EHR; thus making it actionable for patients and their PCPs.

Using a mixed-methods design, this study will be conducted in 2 phases: 1) a formative phase, using the evidence-based user-centered design approach; and 2) a clinical-efficacy phase. For the formative phase, a qualitative research method will be used to: a) adapt MJS to the needs of PCPs and T2D patients; b) integrate MJS DIABETES into the EHR system, the primary care practice and the lives of patients with T2D; and c) evaluate the usability of MJS DIABETES in a subset of T2D patients and their PCPs in order to optimize the tool's performance and workflow integration.

For the clinical efficacy phase, a randomized control trial will be used to identify the efficacy of MJS DIABETES versus Usual Care (UC) on reduction HbA1c at 12-months, among 282 patients with T2D who receive care in safety-net practices.

ELIGIBILITY:
Inclusion Criteria:

Primary Care Provider Inclusion Criteria:

* Fulltime primary care provider (MD/DO, NP) practicing at the participating family health centers (FHCs) and,
* Provide care to at least five patients with a diagnosis of T2D.

Patient Inclusion Criteria:

* Have a diagnosis of T2D for ≥6 months;
* Have uncontrolled T2D defined as HbA1c >7% documented in the EHR on at least two visits in the past year;
* Fluency in English or Spanish;
* Be willing to send/receive text messages; and

Exclusion Criteria:

* Have a diagnosis of T2D for ≥6 months;
* Have uncontrolled T2D defined as HbA1c >7% documented in the EHR on at least two visits in the past year;
* Fluency in English or Spanish;
* Be willing to send/receive text messages; and

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Schoenthaler, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).

REFERENCES:
- [Derived] Mandal S, Belli HM, Cruz J, Mann D, Schoenthaler A. Analyzing User Engagement Within a Patient-Reported Outcomes Texting Tool for Diabetes Management: Engagement Phenotype Study. JMIR Diabetes. 2022 Nov 14;7(4):e41140. doi: 10.2196/41140. PMID 36374531
- [Derived] Schoenthaler A, Cruz J, Payano L, Rosado M, Labbe K, Johnson C, Gonzalez J, Patxot M, Patel S, Leven E, Mann D. Investigation of a Mobile Health Texting Tool for Embedding Patient-Reported Data Into Diabetes Management (i-Matter): Development and Usability Study. JMIR Form Res. 2020 Aug 31;4(8):e18554. doi: 10.2196/18554. PMID 32865505

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: N= 246 participants were enrolled, N=9 of these participants were not randomized to treatment.
Period: Overall Study
Arm/Group | MJS DIABETES | Usual Care
Started | 117 | 120
Completed | 109 | 114
Not Completed | 8 | 6
Not completed — Lost to Follow-up | 1 | 5
Not completed — Withdrawal by Subject | 5 | 1
Not completed — New diagnosis | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MJS DIABETES | Usual Care | Total
Number analyzed (Participants) | 109 | 114 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.54) | 55.7 (9.31) | 56.1 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 66 | 133
  Male | 42 | 48 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 20 | 39
  Not Hispanic or Latino | 90 | 94 | 184
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 38 | 75
  White | 42 | 38 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 30 | 55
Region of Enrollment [Number; unit: participants]
  United States | 109 | 114 | 223

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Level at Baseline
Description: Hemoglobin A1c (HbA1c) extracted from patient medical record. Reported means and 95% confidence intervals are model-adjusted and utilized multiple imputation.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: Percentage of total hemoglobin
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
Percentage of total hemoglobin | 8.37 [8.06 to 8.68] | 8.29 [7.98 to 8.60]

2. Primary Outcome: HbA1c Level at Month 12
Description: as for outcome 1
Time Frame: Month 12
Measure: Mean (95% Confidence Interval); unit: Percentage of total hemoglobin
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
Percentage of total hemoglobin | 8.02 [7.69 to 8.35] | 8.15 [7.82 to 8.48]

3. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Diet Subscale Score
Description: The SDSCA questionnaire is an assessment of diabetes self-management that includes items assessing the following aspects of the diabetes regimen: diet, exercise, blood-glucose testing, and foot care. For each item on the diet subscale, respondents provide the number of days per week (0-7) that they engage in the activity. The total score is the average of all responses and ranges from 0-7; higher scores indicate healthier diet.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.87 (1.68) | 3.42 (1.88)

4. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Diet Subscale Score
Description: as for outcome 3
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.31 (1.64) | 4 (1.84)

5. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Diet Subscale Score
Description: as for outcome 3
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.21 (1.53) | 4.13 (1.65)

6. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Diet Subscale Score
Description: as for outcome 3
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.47 (1.48) | 4.18 (1.67)

7. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Diet Subscale Score
Description: as for outcome 3
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.48 (1.54) | 4.29 (1.66)

8. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Exercise Subscale Score
Description: The SDSCA questionnaire is an assessment of diabetes self-management that includes items assessing the following aspects of the diabetes regimen: diet, exercise, blood-glucose testing and foot care. For each item on the exercise subscale, respondents provide the number of days per week (0-7) that they engage in the activity. The total score is the average of all responses and ranges from 0-7; higher scores indicate greater amounts of exercise.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 2.93 (2.02) | 2.59 (2.07)

9. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Exercise Subscale Score
Description: as for outcome 8
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.56 (2.22) | 2.98 (2.32)

10. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Exercise Subscale Score
Description: as for outcome 8
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.68 (2.1) | 3.1 (2.07)

11. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Exercise Subscale Score
Description: as for outcome 8
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.54 (2) | 3.01 (2.06)

12. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Exercise Subscale Score
Description: as for outcome 8
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.62 (2.09) | 3.26 (2.16)

13. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Blood-Glucose Testing Subscale Score
Description: The SDSCA questionnaire is an assessment of diabetes self-management that includes items assessing the following aspects of the diabetes regimen: diet, exercise, blood-glucose testing and foot care. For each item on the blood-glucose testing subscale, respondents provide the number of days per week (0-7) that they engage in the activity. The total score is the average of all responses and ranges from 0-7; higher scores indicate more frequent weekly blood-glucose testing.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.74 (2.78) | 3.74 (2.9)

14. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Blood-Glucose Testing Subscale Score
Description: as for outcome 13
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.4 (2.79) | 4.07 (2.76)

15. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Blood-Glucose Testing Subscale Score
Description: as for outcome 13
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.32 (2.8) | 3.95 (2.92)

16. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Blood-Glucose Testing Subscale Score
Description: as for outcome 13
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.24 (2.8) | 4.04 (2.87)

17. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Blood-Glucose Testing Subscale Score
Description: as for outcome 13
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.43 (2.71) | 3.98 (2.89)

18. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Foot Care Subscale Score
Description: The SDSCA questionnaire is an assessment of diabetes self-management that includes items assessing the following aspects of the diabetes regimen: diet, exercise, blood-glucose testing and foot care. For each item on the foot care subscale, respondents provide the number of days per week (0-7) that they engage in the activity. The total score is the average of all responses and ranges from 0-7; higher scores indicate more frequent completion of foot care activities.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.12 (2.69) | 3.05 (2.63)

19. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Foot Care Subscale Score
Description: as for outcome 18
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.62 (2.42) | 3.77 (2.54)

20. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Foot Care Subscale Score
Description: as for outcome 18
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.1 (2.58) | 3.89 (2.56)

21. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Foot Care Subscale Score
Description: as for outcome 18
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.27 (2.33) | 3.98 (2.38)

22. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA): Foot Care Subscale Score
Description: as for outcome 18
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.39 (2.29) | 4 (2.4)

23. Secondary Outcome: Michigan Diabetes Knowledge Scale Score
Description: 20-item assessment of diabetes knowledge. Each item has a potential response of "True," "False," and "I don't know." The total score is the number of correct responses normalized by the total number of items responded, and ranges from 0-1; higher scores indicate greater diabetes knowledge.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 0.66 (0.17) | 0.65 (0.14)

24. Secondary Outcome: Michigan Diabetes Knowledge Scale Score
Description: as for outcome 23
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 0.68 (0.16) | 0.64 (0.15)

25. Secondary Outcome: Michigan Diabetes Knowledge Scale Score
Description: as for outcome 23
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 0.71 (0.15) | 0.66 (0.16)

26. Secondary Outcome: Diabetes Self-Efficacy Scale Score
Description: 12-item assessment of participants' confidence in performing certain diabetes-related tasks. For each item, participants select from a Likert scale ranging from 0 (not at all confident) to 10 (very confident). The total score is the sum of responses normalized by the number of items responded and ranges from 0-10; higher scores indicate greater diabetes self-efficacy.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 7.38 (1.86) | 7.42 (1.91)

27. Secondary Outcome: Diabetes Self-Efficacy Scale Score
Description: as for outcome 26
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 7.64 (1.85) | 7.65 (1.86)

28. Secondary Outcome: Diabetes Self-Efficacy Scale Score
Description: as for outcome 26
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 8.09 (1.62) | 7.81 (1.84)

29. Secondary Outcome: Diabetes Self-Efficacy Scale Score
Description: as for outcome 26
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 7.96 (1.58) | 7.49 (2.07)

30. Secondary Outcome: Diabetes Self-Efficacy Scale Score
Description: as for outcome 26
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 8.16 (1.48) | 7.8 (1.78)

31. Secondary Outcome: Interpersonal Processes of Care Score Communication Subscale Score
Description: 18-item assessment of participants' experiences talking with doctors during the study includes items assessing the following aspects of the IPC: 1) Communication, 2) Decision Making, and 3) Inter-personal style. Each item is rated on a Likert scale from 1 (never) to 5 (always). Scores in negative items are reversed. The total scale score is mean of nonmissing items and ranges from 1-5. Higher scores indicate higher frequency of the construct (higher communication scores indicate better patient-provider communication).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.28 (0.71) | 4.34 (0.61)

32. Secondary Outcome: Interpersonal Processes of Care Score Communication Subscale Score
Description: as for outcome 31
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.36 (0.64) | 4.47 (0.58)

33. Secondary Outcome: Interpersonal Processes of Care Score Communication Subscale Score
Description: as for outcome 31
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.31 (0.66) | 4.4 (0.67)

34. Secondary Outcome: Interpersonal Processes of Care Score Communication Subscale Score
Description: as for outcome 31
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.4 (0.61) | 4.49 (0.56)

35. Secondary Outcome: Interpersonal Processes of Care Score Communication Subscale Score
Description: as for outcome 31
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.36 (0.7) | 4.45 (0.55)

36. Secondary Outcome: Interpersonal Processes of Care: Decision Making Subscale Score
Description: 18-item assessment of participants' experiences talking with doctors during the study includes items assessing the following aspects of the IPC: 1) Communication, 2) Decision Making, and 3) Inter-personal style. Each item is rated on a Likert scale from 1 (never) to 5 (always). Scores in negative items were reversed. Total scale score is mean of nonmissing items and ranges from 1-5. Higher scores indicate higher frequency of the construct (higher decision making scores indicate more decision making).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.74 (1.12) | 3.71 (1.14)

37. Secondary Outcome: Interpersonal Processes of Care: Decision Making Subscale Score
Description: as for outcome 36
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.86 (1.01) | 3.97 (1.05)

38. Secondary Outcome: Interpersonal Processes of Care: Decision Making Subscale Score
Description: as for outcome 36
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.93 (1.12) | 3.98 (1.05)

39. Secondary Outcome: Interpersonal Processes of Care: Decision Making Subscale Score
Description: as for outcome 36
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.93 (1.06) | 4.09 (1.02)

40. Secondary Outcome: Interpersonal Processes of Care: Decision Making Subscale Score
Description: as for outcome 36
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 3.93 (1.06) | 4.09 (1.02)

41. Secondary Outcome: Interpersonal Processes of Care: Inter-personal Style Subscale Score
Description: 18-item assessment of participants' experiences talking with doctors during the study includes items assessing the following aspects of the IPC: 1) Communication, 2) Decision Making, and 3) Inter-personal style. Each item is rated on a Likert scale from 1 (never) to 5 (always). Scores in negative items were reversed. Total scale score is mean of nonmissing items and ranges from 1-5. Higher scores indicate higher frequency of the construct (higher inter-personal style scores indicate more inter-personal style).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.48 (0.63) | 4.6 (0.51)

42. Secondary Outcome: Interpersonal Processes of Care: Inter-personal Style Subscale Score
Description: as for outcome 41
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.53 (0.58) | 4.67 (0.5)

43. Secondary Outcome: Interpersonal Processes of Care: Inter-personal Style Subscale Score
Description: as for outcome 41
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.52 (0.56) | 4.61 (0.62)

44. Secondary Outcome: Interpersonal Processes of Care: Inter-personal Style Subscale Score
Description: as for outcome 41
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.47 (0.65) | 4.6 (0.63)

45. Secondary Outcome: Interpersonal Processes of Care: Inter-personal Style Subscale Score
Description: as for outcome 41
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MJS DIABETES | Usual Care
Number analyzed (Participants) | 117 | 120
score on a scale | 4.47 (0.65) | 4.6 (0.63)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | MJS DIABETES | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/120
Other Adverse Events (participants affected / at risk) | 0/117 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT03652389/Prot_SAP_000.pdf